CLINICAL TRIAL: NCT00849511
Title: Melatonin for Migraine Prevention (The MMP-study): A Randomized, Double-blind, Cross-over, Placebo-controlled Study of Melatonin in Prophylactic Treatment of Migraine
Brief Title: Melatonin for Migraine Prevention
Acronym: MMP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nordlandssykehuset HF (Other)
Collaborators: University of Tromso (Other)
Responsible Party: Principal Investigator, Karl B. Alstadhaug, MD, PhD, Nordlandssykehuset HF
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 270472
Record Dates: First submitted 2009-02-23; First posted 2009-02-24 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Migraine
Keywords: Migraine prevention; Crossover; Melatonin
MeSH Terms: conditions — Migraine Disorders | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo first (Active Comparator): Placebo 8 weeks, 6 weeks washout, extended-release melatonin 2 mg vesper for 8 weeks
  Interventions: Drug: melatonin
- Melatonin first (Active Comparator): Extended-release melatonin 2 mg vesper for 8 weeks, 6 weeks washout, placebo 8 weeks
  Interventions: Drug: melatonin

INTERVENTIONS:
Drug: melatonin — Circadin (melatonin) 2 mg ret. TAB vesp. for 8 weeks
  Other Names: Circadin

SUMMARY:
The circadian system with its centre in the hypothalamus is involved in migraine pathophysiology. Whether it plays a pivotal role is not clarified. The investigators postulate that a destabilized circadian system may increase migraine attack susceptibility, and that stabilization by supplying melatonin a migraine preventive effect will be achieved.

A previous open label study has shown effects that certainly warrant a placebo controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 65 years, both male and females.
* Migraine present for at least 1 year and fulfilling diagnostic criteria that conform to those of the International Headache Society (HIS) [2] but otherwise healthy.
* Attacks of migraine should occur 4-6 times per month, there should be no regular use of other drugs, and the patient has to be able to differentiate between migraine headache and non-migrainous headache.
* Preventive drugs for migraine should not have been used the last three months.
* Conventional acute attack treatment is accepted, but not sporadic use of other drugs like hypnotics and anxiolytics.
* Residence of North-Norway.

Exclusion Criteria:

* Medication overuse headache, chronic migraine.
* Pregnant and breast feeding women.
* Patient with either serious co-morbidity or conditions requiring medical treatment or caution.
* Psychiatric disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-02; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Migraine attack frequency | 8 weeks

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index score | 8 weeks
Night time sleep quality | 8 weeks
Point prevalence of insomnia | 8 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Departement of Neurology, NLSH HF, Bodø
  - Departement of Neurology, Tromsø

REFERENCES:
- [Background] Peres MF, Zukerman E, da Cunha Tanuri F, Moreira FR, Cipolla-Neto J. Melatonin, 3 mg, is effective for migraine prevention. Neurology. 2004 Aug 24;63(4):757. doi: 10.1212/01.wnl.0000134653.35587.24. No abstract available. PMID 15326268